CLINICAL TRIAL: NCT00462891
Title: Breast Cancer Screening and Follow-Up in a PBRN: The Mammography FastTrack Trial
Brief Title: A Mammography FastTrack Program in Increasing the Number of Women Undergoing Breast Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael J. Barry, MD, Project Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 02-114; R21CA121908 (NIH); MGH-2005-P-002474/1
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IT System (Experimental): IT system to send reminder letters to patients overdue for breast cancer screening.
  Interventions: Other: IT System
- Usual Care (No Intervention)

INTERVENTIONS:
Other: IT System
  Arms: IT System

SUMMARY:
RATIONALE: Screening may help doctors find breast cancer cells early and plan better treatment for breast cancer. The Mammography FastTrack program may be effective in increasing the number of patients who undergo mammography.

PURPOSE: This randomized clinical trial is studying the use of a Mammography FastTrack program to increase the number of women who undergo mammography.

DETAILED DESCRIPTION:
OBJECTIVES:

* Classify all patients within the Massachusetts General Primary Care-Practice Based Research Network (MGPC-PBRN) according to patient-primary care provider (PCP) linkage status.
* Develop a breast cancer screening intervention program called Mammography FastTrack that facilitates the ordering of mammograms to be used either by PCPs (for PCP-linked patients) or by practice managers (for practice-linked patients).
* Compare the impact of the Mammography FastTrack program on mammography screening rates in PCP-linked vs practice-linked patients overdue for breast cancer screening.

OUTLINE: This is a randomized, multicenter study.

Mammography-eligible women are linked to either a provider or a practice within the Massachusetts General Primary Care Practice-Based Research Network (MGPC-PBRN). Practices within the MGPC-PBRN are stratified according to baseline mammography screening rates (high vs low) and practice type (community health center vs hospital-based vs community-based) and are randomized to 1 of 2 arms.

* Arm I: Physicians and practice managers receive e-mail alerts at months 1 and 3 informing them of the availability of mammography screening data for their panel of primary-care patients. A hyperlink refers the provider to a web-portal for the Mammography FastTrack program that lists all eligible patients who have not undergone mammography. The provider may then click a button to schedule, defer (providing reason for deferral), or provide the date of a recent mammogram.
* Arm II: Practices continue standard care. At the end of 12 months, electronic report and billing data and a review of electronic health records are used to determine the completion of mammograms.

PROJECTED ACCRUAL: A total of 6,730 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Any outpatient at a participating Massachusetts General Primary Care Practice-Based Research Network (MGPC-PBRN) practice within the past 3 years

  * No patient who the Massachusetts General Hospital system lists as having a primary care provider who is not in one of the MGPC-PBRN networks (linking patients with a provider or practice)
  * No patient who is not linked to specific provider or practice (randomized portion of study)
* Billing, scheduling, and clinical electronic data sources required
* No mammogram within the past 2 years (randomized portion of study)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Age 42 to 69 years (randomized portion of study)
* Female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* No prior bilateral mastectomy (randomized portion of study)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6730 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Proportion of overdue patients completing mammography screening in intervention and control groups | 1 year
  Proportion of overdue patients completing mammography screening in intervention and control groups over the 1-year study.

SECONDARY OUTCOMES:
Difference in percentage of patients overdue at baseline receiving mammogram during the study period in intervention and control practices at 6 months | 1 year
Comparison of time to mammography completion in intervention vs control groups | 1 year
Clinical and nonclinical outcomes recorded by Mammography FastTrack tool | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Barry, MD, Study Chair — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Atlas SJ, Grant RW, Lester WT, Ashburner JM, Chang Y, Barry MJ, Chueh HC. A cluster-randomized trial of a primary care informatics-based system for breast cancer screening. J Gen Intern Med. 2011 Feb;26(2):154-61. doi: 10.1007/s11606-010-1500-0. Epub 2010 Sep 15. PMID 20872083
- [Derived] Atlas SJ, Ashburner JM, Chang Y, Lester WT, Barry MJ, Grant RW. Population-based breast cancer screening in a primary care network. Am J Manag Care. 2012 Dec;18(12):821-9. PMID 23286611